CLINICAL TRIAL: NCT06896097
Title: Ridge Preservation Using Collagen Sponge Alone or Combined with Xenograft: a Clinical and Histological Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Zeinab Shalaby, lecturer of oral medicine, periodontology, diagnosis and radiology Department faculty of Dental Medicine Al-Azhar University, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: P-ME-21-06
Record Dates: First submitted 2022-08-24; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Ridge Preservation

STUDY DESIGN:
Intervention Model Description: The design of this clinical trial will be randomized double blind technique; the randomization of the patients will be performed through a computer program, patients will be subjected to extraction of primary maxillary single rooted tooth and socket preservation will be done by collagen sponge alone or combined with xenograft
Who Masked: Participant
Masking Description: The design of this clinical trial will be randomized double blind technique; the randomization of the patients will be performed through a computer program
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (Experimental): including 8 patients, preservation of extraction sockets will be done with combination of collagen sponge (deep collagen layer) and xenograft will be placed on top of the collagen sponge to fill the coronal part of the socket and socket sealing will be performed with a new layer of collagen sponge (superficial collagen layer) and criss-cross suture to stabilize the graft in place
  Interventions: Procedure: Ridge preservation
- Group II (Experimental): including 8 patients, preservation of extraction sockets will be done with collagen spong alone and criss-cross suture
  Interventions: Procedure: Ridge preservation
- Group III (Experimental): control group, including 8 patients, preservation of extraction sockets will be done with atraumatic extraction and left for spontaneous healing with criss -cross suture
  Interventions: Procedure: Ridge preservation

INTERVENTIONS:
Procedure: Ridge preservation — extraction of non restorable tooth in a traumatic way and socket preservation with the selected group

SUMMARY:
24 patients had a treatment plan for extraction of non restorable single rooted maxillary tooth and will be subjected to one of three groups after tooth extraction Group (I): including 8 patients, preservation of extraction sockets will be done with combination of collagen sponge and xenograft will be placed on top of the collagen sponge to fill the coronal part of the socket, till crestal bone level and socket sealing will be done with a new layer of collagen sponge(superficial collagen layer) and criss-cross suture to stabilize the graft in place.

Group (II): including 8 patients, preservation of extraction sockets will be done with collagen sponge alone and criss-cross suture. Group (III): control group, including 8 patients, preservation of extraction sockets will be done with atraumatic extraction and left for spontaneous healing with criss-cross suture.

DETAILED DESCRIPTION:
- Surgical Phase:

* Local infiltration anesthesia will be first administered to all patients in this study.
* Teeth will be extracted, using a flapless approach a traumatically as much as possible.
* Atraumatic extraction will start with dissection of periodontal ligaments in crestal part using 15C blades mounted over a round-handed blade to facilitate rotation without lacerating the soft tissue
* Then teeth will be luxated using micro-elevators and the final delivery movement will be done using forceps.
* Sockets will be thoroughly debrided using a curette, especially in case with periapical lesions, to ensure complete removal of granulation tissue.
* Assessment of sockets walls integrity will be done visually and using a UNC-15 periodontal probe. All patients will be allocated into one of the three study groups. Group (I): including 8 patients, preservation of extraction sockets will be done with combination of collagen sponge and xenograft will be placed on top of the collagen sponge to fill the coronal part of the socket, till crestal bone level and socket sealing will be done with a new layer of collagen sponge(superficial collagen layer) and criss-cross suture to stabilize the graft in place.

Group (II): including 8 patients, preservation of extraction sockets will be done with collagen sponge and criss-cross suture. Group (III): control group, including 8 patients, preservation of extraction sockets will be done with atraumatic extraction and left for spontaneous healing with criss-cross suture.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a single rooted maxillary tooth that had a treatment plan of extraction as; endodontic complication, root fracture, trauma, or advanced carious lesions.
* Teeth with or without periapical lesions not affecting buccal wall integrity.
* Patients age (18 - 60) years old.
* Patients with clinical periodontal health on an intact periodontium and adequate volume that allow for implant placement after follow-up period.
* Pristine extraction socket (type I socket).

Exclusion Criteria:

* Patients with any systemic condition that may affect surgical and healing process.
* Patients with active acute infection related to teeth of interest.
* Pregnant females.
* History of malignancy or radiotherapy for malignancy in the past 5 years.
* History of active bone metabolic disease.
* Patients taking or were taking medications that may affect bone turnover such as bisphosphonates.
* Patients with buccal bone thickness less than 1 mm that necessitate regeneration and flap elevation. 7
* Smoker patients who reported tobacco use in the past 5 years.
* The design of this clinical trial will be randomized double blind technique; the randomization of the patients will be performed through a computer program.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Ridge preservation using collagen sponge alone or combined with xenograft clinical and histological | 4 months
  evaluate and compare the clinical outcomes to width and height of socket preservation using the Biologically-oriented Alveolar Ridge Preservation (BARP) versus Collagen Sponge (CS), all compared to negative control

CONTACTS AND LOCATIONS:
Overall Officials: Zienab Shalaby, Principal Investigator — Faculty of Dental Medicine for Girls
Locations (1):
- Faculty of Dental Medicine for Girls, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No